CLINICAL TRIAL: NCT04969913
Title: Community Dynamics of Malaria Transmission in Humans and Mosquitoes at Maferinyah Sub-prefecture, Guinea
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000160; 000160-I
Record Dates: First submitted 2021-07-20; First posted 2021-07-21 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Malaria
Keywords: Assays; BLOOD SAMPLING; Parasites; Gametocytes; Infection; Natural History
MeSH Terms: conditions — Malaria; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 19 + years: Healthy adults over the age of 19 years
- Ages 11 - 18 years: Healthy children between the ages of 11 and 18 years
- Ages 5 - 10 years: Healthy children between the ages of 5 and 10 years
- Ages 6 months - 4 years: Healthy infants between the ages of 6 months and four years

SUMMARY:
Background:

Half of the world s population is at risk of malaria. In 2015, there were 214 million cases of malaria and 438,000 deaths. A transmission-blocking vaccine (TBV) could help end the disease. Improved tests are needed to measure how well the vaccines work. Researchers want to collect data about malaria infection as the first step in testing a TBV in rural Guinea.

Objective:

To study community dynamics of malaria transmission by estimating the rate of blood smear positive people by month and season.

Eligibility:

People 6 months of age and older who live in Maf(SqrRoot)(Registered Trademark)rinyah sub-prefecture and plan to remain during the study. Households with at least 3 people who are eligible to take part in the study are also needed.

Design:

Participants will be screened with a medical and medicine history. They will have a physical exam. Their height and weight will be measured. Their vital signs may be taken.

Participants will have a study visit each month for up to 3 years. They will get a study ID. They will be asked about any symptoms of malaria or changes in health. They will give blood samples. They may have a physical exam. Within 3 days of the study visits, live and dead mosquitoes may be gathered in and around their home. Insecticide spray will be used.

Participants can visit the clinic at any time if they feel ill. If they have malaria, they will be treated according to Guinea National Malaria Control Guidelines for adults and children.

DETAILED DESCRIPTION:
A vaccine that interrupts malaria transmission is critical to eradicate the disease, but improved assays are needed to measure the efficacy of vaccines. Transmission-blocking vaccines (TBVs) work by inducing antibodies that inhibit parasite development in the mosquito interrupting transmission. Efficacy of vaccines may be estimated by in vitro membrane feeding assays using immune sera and laboratory mosquitoes, but qualified assays that measure transmission in the field are needed to assess transmission-blocking interventions in natura.

Clinical trials of TBVs have started elsewhere on the continent in Mali, and we expect to expand TBV studies in Guinea in the near future. This protocol will use a longitudinal cohort to gather information of malaria transmission based on the rates of blood smear positive individuals by month, season and year in at Maferinyah sub-prefecture, Guinea.

Individuals in the villages will be approached first for participation, including permission to contact their household and neighbors of their compound for participation. Households will be identified using census data and individuals will be consented for participation.

Malaria smears will be obtained at monthly visits, in conjunction with mosquito collections in/around village residences. Parasite infection rates in locally caught mosquitoes will be assessed longitudinally for differences by season and year. A total of 400 volunteers from Maferinyah will be enrolled. Participants will be followed for up to 3 years, to collect data that will guide the design of future community-based trials of TBV.

ELIGIBILITY:
* SUBJECT INCLUSION CRITERIA:
* 6 months of age and above
* Known resident of Maferinyah sub-prefecture and planning to remain for duration of study
* Willingness to allow stored laboratory specimens to be used for future research
* Acceptance and signature of the written informed consent and the assent for children aged 12-17 years who are not otherwise emancipated

HOUSEHOLD INCLUSION CRITERIA:

To be eligible for participation, households must meet the following criteria:

* Household with at least 3 residents eligible for participation.
* Household with at least one compound member who is below 18 years of age whose parents or caretakers are willing to provide informed consent for the child to participate
* Household members willing to accommodate mosquito sampling in their compound, both indoors and outdoors.

SUBJECT EXCLUSION CRITERIA:

* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the subject to understand and cooperate with the study protocol.
* Other condition that, in the opinion of the investigator, would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy Guinean infants, children, and adults (any age) from Maferinyah sub-prefecture. Maferinyah is a town and sub-prefecture in the Forecariah Prefecture in the Kindia Region of western Guinea. Maferinyah is located about 50 kms directly to the west (and 75 kms by paved road) of Conakry, the capital city of Guinea
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2024-10-23 (Actual)

PRIMARY OUTCOMES:
To study community dynamics of malaria transmission by estimating the rate of blood smear positive individuals by month and season stratified by age | Season and year
  Rate of blood smear positive individuals by month and season stratified by age

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer C Hume, Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- Immunology and Pathogenesis Laboratories, Bethesda, Maryland, United States
- Maferinyah Rural Health Training and Research Center, Maferinyah, Guinea

IPD SHARING:
Plan to Share IPD: No